CLINICAL TRIAL: NCT01746394
Title: Delta Healthy Sprouts: A Randomized Trial to Determine the Comparative Efficacy of Two Maternal, Infant, and Early Childhood Home Visiting Programs on Maternal Weight Control and Childhood Obesity in the Mississippi Delta
Brief Title: Delta Healthy Sprouts: Intervention to Promote Maternal Weight Control and Reduce Childhood Obesity in the MS Delta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Delta Human Nutrition Research Program (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DHN_12_01
Record Dates: First submitted 2012-12-05; First posted 2012-12-10 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-02

CONDITIONS: Obesity
Keywords: obesity; pregnant women; nutrition assessment; health behavior
MeSH Terms: conditions — Obesity; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parents as Teachers Enhanced (Experimental): Participants in the Parents as Teachers Enhanced (PaTE) intervention arm will receive the enhanced diet and activity maternal, infant, and early childhood home visiting program
  Interventions: Behavioral: Parents as Teachers Enhanced; Behavioral: Parents as Teachers
- Parents as Teachers (Active Comparator): Participants in the Parents as Teachers (PaT) control arm will receive the standard maternal, infant, and early childhood home visiting program
  Interventions: Behavioral: Parents as Teachers

INTERVENTIONS:
Behavioral: Parents as Teachers Enhanced — Participants will receive the same monthly Parents as Teachers (PaT) lessons and materials at each home visit as the PaT arm. Additionally, these mothers will receive the enhanced nutrition and physical activity lessons and materials which will follow the family well-being format of the PaT lessons. The StartSmart lessons will focus on healthy gestational weight gain, diet, physical activity, breastfeeding, weight management, healthy eating, food shopping, meal preparation, physical activity, proper infant feeding, and infant activity time.
  Other Names: PaTE
  Arms: Parents as Teachers Enhanced
Behavioral: Parents as Teachers — Participants will receive monthly Parents as Teachers (PaT) lessons and materials at each home visit. The Parent Educator will first connect with the mother by discussing or reviewing content from the prior visit; reflect on the mother's experience with continuing the parent-child activity from the prior visit; and agree on what will happen during the current visit. For the lesson plan, the Parent Educator will cover the following three areas using discussion, activities, and handouts: parent-child interaction, develop-centered parenting, and family well-being. In closing, the Parent Educator will review and evaluate the visit, talk about the mother's next step, and plan for the next visit.
  Other Names: PaT

SUMMARY:
The Delta Healthy Sprouts Project is a randomized, controlled trial evaluating the enhancement of an existing Mother, Infant, and Early Childhood Home Visiting Program in 150 African American women in their early second trimester of pregnancy. The control arm, Parents as Teachers, is an evidence-based approach to increase parental knowledge of child development and improve parenting practices. The experimental arm, Parents as Teachers Enhanced, builds on the Parents as Teachers curriculum by including nutrition and physical activity components specifically designed for the gestational and postnatal periods. Both arms of the intervention will be implemented by community-based, trained Parent Educators. The comparative effectiveness of the two intervention arms on weight status, dietary intake, and health behaviors of mothers and their infants will be assessed. The Delta Healthy Sprouts Project will determine if a novel, scalable, lifestyle intervention can improve the health of African American women and their children at high-risk for obesity and chronic disease.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Less than 18 weeks pregnant with first, second, or third child
* Resident of Mississippi counties of Washington and Bolivar

Exclusion Criteria:

* Pregnant with more than one fetus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Gestational weight gain | 9 months gestation
  Percentages of gestational weight gain which fall within the ranges recommended by the Institute of Medicine (based on pre-pregnancy body mass index)
Maternal postpartum weight retention | 12 months postnatal
  Amount of weight retained at 12 months postpartum compared to self-reported pre-pregnancy weight
Maternal dietary intake | 12 months postpartum
  Dietary intake measured using 24-hour dietary recall
Maternal physical activity | 12 months postpartum
  Physical activity measured using a physical activity questionnaire
Infant dietary intake | 12 months after birth
  Dietary intake measured using 24-hour dietary recall as reported by mother
Infant activity | 12 months after birth
  Activity measured using responses to questions concerning time spent confined (e.g. in infant seat) and unconfined (e.g. on play mat)
Infant body mass index | 12 months after birth
  Incremental body mass index during the first year of life

SECONDARY OUTCOMES:
Breastfeeding | 12 months postpartum
  Breastfeeding initiation and continuation for first 12 months after birth of infant
Home food environment | 12 months postpartum
  Measured using home food inventory; based on direct observation of foods in household (i.e. in refrigerator, freezer, pantry, cupboards, or other areas food is stored)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Thomson, PhD, Principal Investigator — USDA Agricultural Research Service; Lisa M Tussing-Humphreys, PhD, Study Chair — University of Illinois at Chicago
Locations (1):
- USDA Agricultural Research Service Mid South Area Office, Stoneville, Mississippi, United States

REFERENCES:
- [Background] Thomson JL, Tussing-Humphreys LM, Goodman MH. Delta Healthy Sprouts: a randomized comparative effectiveness trial to promote maternal weight control and reduce childhood obesity in the Mississippi Delta. Contemp Clin Trials. 2014 May;38(1):82-91. doi: 10.1016/j.cct.2014.03.004. Epub 2014 Mar 29. PMID 24685997
- [Derived] Thomson JL, Tussing-Humphreys LM, Goodman MH, Landry AS. Infant activity and sleep behaviors in a maternal and infant home visiting project among rural, southern, African American women. Matern Health Neonatol Perinatol. 2018 May 16;4:10. doi: 10.1186/s40748-018-0078-0. eCollection 2018. PMID 29785275
- [Derived] Thomson JL, Tussing-Humphreys LM, Landry AS, Goodman MH. No Improvements in Postnatal Dietary Outcomes Were Observed in a Two-Arm, Randomized, Controlled, Comparative Impact Trial among Rural, Southern, African-American Women. J Acad Nutr Diet. 2018 Jul;118(7):1196-1207. doi: 10.1016/j.jand.2017.11.010. Epub 2018 Feb 1. PMID 29396153
- [Derived] Tussing-Humphreys LM, Thomson JL, Hemphill NO, Goodman MH, Landry AS. Maternal weight in the postpartum: results from the Delta healthy sprouts trial. Matern Health Neonatol Perinatol. 2017 Dec 4;3:20. doi: 10.1186/s40748-017-0058-9. eCollection 2017. PMID 29214042
- [Derived] Thomson JL, Tussing-Humphreys LM, Goodman MH, Landry AS, Olender SE. Low rate of initiation and short duration of breastfeeding in a maternal and infant home visiting project targeting rural, Southern, African American women. Int Breastfeed J. 2017 Apr 8;12:15. doi: 10.1186/s13006-017-0108-y. eCollection 2016. PMID 28405211
- [Derived] Thomson JL, Tussing-Humphreys LM, Goodman MH, Olender SE. Physical Activity Changes during Pregnancy in a Comparative Impact Trial. Am J Health Behav. 2016 Nov;40(6):685-696. doi: 10.5993/AJHB.40.6.1. PMID 27779937
- [Derived] Thomson JL, Tussing-Humphreys LM, Goodman MH, Olender SE. Gestational Weight Gain: Results from the Delta Healthy Sprouts Comparative Impact Trial. J Pregnancy. 2016;2016:5703607. doi: 10.1155/2016/5703607. Epub 2016 Aug 9. PMID 27595023
- [Derived] Tussing-Humphreys LM, Thomson JL, Goodman MH, Olender S. Maternal diet quality and nutrient intake in the gestational period: results from the delta healthy sprouts comparative impact trial. Matern Health Neonatol Perinatol. 2016 Aug 17;2:8. doi: 10.1186/s40748-016-0036-7. eCollection 2016. PMID 27536380